CLINICAL TRIAL: NCT00034307
Title: A Randomized, Double-Blind, Placebo-Controlled Safety and Efficacy Study of Sitaxsentan Sodium Treatment in Patients With Pulmonary Arterial Hypertension
Brief Title: Safety and Efficacy of Sitaxsentan in the Treatment of Pulmonary Arterial Hypertension
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ICOS-Texas Biotechnology (Industry)
Collaborators: ICOS Corporation (Industry); Texas Biotechnology Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FPH01/FPH01-X
Record Dates: First submitted 2002-04-24; First posted 2002-04-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-05

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

INTERVENTIONS:
Drug: sitaxsentan sodium

SUMMARY:
This is a clinical research study designed to evaluate an investigational new medication called sitaxsentan for the treatment of pulmonary arterial hypertension (patients with NYHA functional class II, III or IV). The purpose of this study is to evaluate the safety and effectiveness of two different doses of sitaxsentan, compared to placebo (inactive treatment) for the treatment of pulmonary arterial hypertension. Patients who complete this trial may be eligible to take part in an extension trial (Protocol FPH01-X). Eligible patients who receive placebo in the 12-week study cross over to receive sitaxsentan for the extension trial.

ELIGIBILITY:
Inclusion Criteria:

1. NYHA Class II, III or IV
2. 16 to 75 years of age
3. Specific peak VO2 range
4. PPH, PAH due to connective tissue disease or select congenital heart disease
5. Qualifying cardiac catheterization
6. History of CXR and qualifying pulmonary function test
7. History of qualifying ventilation-perfusion lung scan
8. History of qualifying echocardiogram
9. Women of childbearing potential must use contraceptives
10. Stable dose of corticosteroids if prescribed

Exclusion Criteria:

1. Significant lung disease
2. Chronic liver disease
3. Uncontrolled sleep apnea
4. History of specific types of left heart disease
5. Any disorder that compromises ability to give informed consent
6. Uncontrolled sleep apnea
7. Inability to perform bicycle exercise test
8. On-going treatment with an experimental drug or device within the last 30 days
9. HIV infection
10. Specific liver dysfunction
11. Chronic renal disease
12. Pregnancy/Nursing
13. Chronic active hepatitis B or C
14. Chronic Flolan or Tracleer use within the last 30 days

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180

CONTACTS AND LOCATIONS:
Overall Officials: Lyn Frumkin, M.D., Ph.D., Study Director — ICOS Corporation
Locations (26):
- United States (25):
  - University of Southern California Hospital, Ambulatory Health Sciences, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Harbor-UCLA Medical Center, Torrance, California
  - The Children's Hospital, Denver, Colorado
  - University of Colorado/ Health Science Center, Denver, Colorado
  - Emory University Hospital - McKelvey Lung Transplantation Center, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Rush Heart Institute, Center for Pulmonary Heart Disease, Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - LSU - School of Medicine, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan Hospital, Division of Cardiology, Ann Arbor, Michigan
  - Mayo Clinic - Division of Cardiovascular Disease, Rochester, Minnesota
  - Columbia Presbyterian Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic Foundation, Department of Pulmonary and Critical Care, Cleveland, Ohio
  - Division of Cardiology - The Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health Sciences, Portland, Oregon
  - University of Pittsburgh Medical Center, CHF/Transplantation Cardiology, Pittsburgh, Pennsylvania
  - Pulmonary Division - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine Pulmonary & Critical Care Section, Houston, Texas
  - University of Wisconsin Medical School, Milwaukee, Wisconsin
- SMBD Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- See also: Pulmonary Hypertension Association — http://www.phassociation.org